CLINICAL TRIAL: NCT05969223
Title: A Phase 4 Multicenter, Randomized, Double-Blind Study of Risankizumab for the Treatment of Adult Subjects With Moderate to Severe Genital Psoriasis or Moderate to Severe Scalp Psoriasis
Brief Title: Study to Assess the Safety and Efficacy of Subcutaneously Injected Risankizumab in Adult Participants With Genital or Scalp Psoriasis
Acronym: UnlIMMited
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M23-702; 2023-504154-35-00 (Other: EU CT)
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Genital Psoriasis; Scalp Psoriasis
Keywords: Genital Psoriasis; Scalp Psoriasis; Plaque Psoriasis; Psoriasis; ABBV066; Skyrizi; Risankizumab
MeSH Terms: conditions — Psoriasis | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Study-G Placebo (Period A) (Placebo Comparator): Participants with moderate to severe genital psoriasis received placebo for risankizumab subcutaneously at Weeks 0 and 4 during Period A.
  Interventions: Drug: Placebo for Risankizumab
- Study-G Risankizumab (Period A) (Experimental): Participants with moderate to severe genital psoriasis received 150 mg of risankizumab subcutaneously at Weeks 0 and 4 during Period A.
  Interventions: Drug: Risankizumab
- Study-S Placebo (Period A) (Placebo Comparator): Participants with moderate to severe scalp psoriasis received placebo for risankizumab subcutaneously at Weeks 0 and 4 during Period A.
  Interventions: Drug: Placebo for Risankizumab
- Study-S Risankizumab (Period A) (Experimental): Participants with moderate to severe scalp psoriasis received 150 mg of risankizumab subcutaneously at Weeks 0 and 4 during Period A.
  Interventions: Drug: Risankizumab
- Study-G Placebo/Risankizumab (Period B) (Experimental): Participants with moderate to severe genital psoriasis received placebo for risankizumab during Period A, and 150 mg of risankizumab subcutaneously at Weeks 16, 28, and 40 during Period B.
  Interventions: Drug: Risankizumab
- Study-G Risankizumab/Risankizumab (Period B) (Experimental): Participants with moderate to severe genital psoriasis received 150 mg of risankizumab subcutaneously during Period A, and continued with this treatment at Weeks 16, 28, and 40 during Period B.
  Interventions: Drug: Risankizumab
- Study-S Placebo/Risankizumab (Period B) (Experimental): Participants with moderate to severe scalp psoriasis received placebo for risankizumab during Period A, and 150 mg of risankizumab subcutaneously at Weeks 16, 28, and 40 during Period B.
  Interventions: Drug: Risankizumab
- Study-S Risankizumab/Risankizumab (Period B) (Experimental): Participants with moderate to severe scalp psoriasis received 150 mg of risankizumab subcutaneously during Period A, and continued with this treatment at Weeks 16, 28, and 40 during Period B.
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Risankizumab — Subcutaneous injection
  Other Names: Skyrizi; ABBV-066
  Arms: Study-G Placebo/Risankizumab (Period B); Study-G Risankizumab (Period A); Study-G Risankizumab/Risankizumab (Period B); Study-S Placebo/Risankizumab (Period B); Study-S Risankizumab (Period A); Study-S Risankizumab/Risankizumab (Period B)
Drug: Placebo for Risankizumab — Subcutaneous injection
  Arms: Study-G Placebo (Period A); Study-S Placebo (Period A)

SUMMARY:
Psoriasis (PsO) is a chronic disease characterized by marked inflammation of the skin that results in thick, red, scaly plaques. This study will assess how safe and effective risankizumab is in adult participants with moderate to severe genital psoriasis or moderate to severe scalp psoriasis. Adverse events and change in disease signs and symptoms will be monitored.

Risankizumab (Skyrizi) is a drug being studied for the treatment of moderate to severe genital psoriasis or moderate to severe scalp psoriasis. Approximately 200 participants with moderate to severe genital psoriasis or moderate to severe scalp psoriasis will be enrolled across approximately 45 sites globally.

The study will be broken up into 2 studies by disease location, participants with moderate to severe genital psoriasis (Study-G) and moderate to severe scalp psoriasis (Study-S). In both studies participants will receive subcutaneous (SC) injections of risankizumab during the 52 week treatment period, or SC injections of placebo risankizumab during the 16 week treatment period followed by SC injections of risankizumab during the 36 week treatment period, with an 8-week follow-up period after the 52 week treatment period.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

DETAILED DESCRIPTION:
Safety and efficacy data through 22 January 2025 are included in the interim analysis, which was conducted after all participants completed Week 16 of Study-G or Study-S in Period A.

ELIGIBILITY:
Inclusion Criteria:

* Must have clinical diagnosis of chronic plaque psoriasis with or without psoriatic arthritis for at least 6 months before the baseline visit.
* Must have a current diagnosis of moderate to severe genital psoriasis (Study-G) defined as static Physician Global Assessment of Genitalia (sPGA-G) ≥ 3 or moderate to severe scalp psoriasis (Study-S) defined as Psoriasis Scalp Severity Index (PSSI) >= 12, scalp Investigator Global Assessment (IGA) >= 3, and >= 30% of the scalp affected.
* Must have body surface area (BSA) ≥ 1% with at least 60% of subjects having BSA ≥ 10%; sPGA ≥ 3; inadequate control of psoriasis and/or intolerance to topical treatment, phototherapy and/or systemic therapy; and be candidates for systemic therapy or phototherapy as assessed by the investigator.

Exclusion Criteria:

* Had previous exposure to IL-23 inhibitors including but not limited to guselkumab, tildrakizumab, ustekinumab, mirikizumab, or risankizumab.
* History of an allergic reaction or significant sensitivity to constituents of the study drug (and its excipients) and/or other products in the same class.
* Non-plaque forms of psoriasis or other active skin disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
Study-G: Percentage of Participants with Achievement of static Physician Global Assessment of Genitalia (sPGA-G) of 0 or 1 | Week 16
  The sPGA-G is a 6-point score ranging from 0 to 5, with a larger score indicating greater severity, based on the physician's assessment of the average thickness, erythema, and scaling of psoriatic genital lesions.
Study-S: Percentage of Participants with Achievement of Scalp Investigator Global Assessment (IGA) of 0 or 1 | Week 16
  The scalp IGA is a measurement of overall scalp involvement by the investigator at the time of evaluation. The scalp IGA is a 5-point scale ranging from 0 (clear) to 4 (severe) incorporating an assessment of the severity of the 3 primary signs of the disease: erythema, scaling, and plaque elevation.

SECONDARY OUTCOMES:
Study-G: Percentage of Participants with Achievement of static Physician Global Assessment of Genitalia (sPGA-G) of 0 | Week 16
  The sPGA-G is a 6-point score ranging from 0 to 5, with a larger score indicating greater severity, based on the physician's assessment of the average thickness, erythema, and scaling of all psoriatic lesions.
Study-G: Percentage of Participants with Achievement of Dermatology Life Quality Index (DLQI) of 0 or 1 | Week 16
  The DLQI is a self-administered, 10-question questionnaire covering 6 domains (symptoms and feelings, daily activities, leisure, work and school, personal relationships, treatment) and has a 1-week recall period. The response options range from 0 (not affected at all) to 3 (very much affected). This gives an overall range of 0 to 30 where lower scores mean better quality of life.
Study-G: Percentage of Participants with Achievement of Clinically Meaningful (>= 4-point) Improvement from Baseline on the Genital Psoriasis Itch Numerical Rating Scale (NRS) [Among Participants with a Baseline Score >= 4] | Week 16
  The scalp Itch NRS is a self-administered NRS that asks the patients to assess their scalp itch on a scale from 0 to 10 where 0 represents no itch and 10 represents worst imaginable itch.
Study-G: Percentage of Participants with Achievement of Genital Psoriasis Sexual Frequency Questionnaire (GenPs-SFQ) Item 2 score of 0 or 1 Among Participants with a Baseline score >= 2 | Week 16
  The GenPs-SFQ is a patient-reported outcome(s) [PRO] measure to evaluate the impact of genital psoriasis symptoms on sexual frequency, using a 1-week recall period. It consists of 2 items that assess the impact of genital psoriasis symptoms on the frequency of sexual activity. Each item uses a Likert scale. Respondents are asked to answer the questions based on their psoriasis symptoms in the genital area. Genital area is defined as the labia majora (outer lip), labia minora (inner lip), and perineum (area between vagina and anus) for females; penis, scrotum, and perineum (area between the penis and anus) for males.
Study-S: Percentage of Participants with Achievement of Psoriasis Scalp Severity Index (PSSI 90) | Week 16
  PPSI 90 is defined as >= 90% improvement from baseline in PSSI. The physician will assess the severity of scalp psoriasis using the PSSI, which consists of an assessment of erythema, induration, and desquamation on a scale from 0 (none) to 4 (very severe) and the percentage of scalp involved on a scale from 1 (<10% of scalp involved) to 6 (90 to 100% of scalp involved). The composite score is calculated as the sum of the scores for erythema, induration and desquamation multiplied by the score recorded for the extent of scalp area involved. The PSSI ranges from 0 to 72.
Study-S: Percentage of Participants with Achievement of PSSI 75 | Week 16
  PPSI 75 is defined as >= 75% improvement from baseline in PSSI. The physician will assess the severity of scalp psoriasis using the PSSI, which consists of an assessment of erythema, induration, and desquamation on a scale from 0 (none) to 4 (very severe) and the percentage of scalp involved on a scale from 1 (<10% of scalp involved) to 6 (90 to 100% of scalp involved). The composite score is calculated as the sum of the scores for erythema, induration and desquamation multiplied by the score recorded for the extent of scalp area involved. The PSSI ranges from 0 to 72.
Study-S: Change from Baseline in Psoriasis Symptom Scale (PSS) | Week 16
  The PSS is a 4-item PRO instrument that assesses the severity of psoriasis symptoms in patients with moderate to severe psoriasis, using a recall period of 1 day. The symptoms include pain, redness, itching and burning from psoriasis. Current symptom severity is assessed using a 5-point Likert-type scale ranging from 0 (none) to 4 (very severe).
Study-S: Percentage of Participants with Achievement of PSSI 100 | Week 16
  PPSI 100 is defined as >= 100% improvement from baseline in PSSI. The physician will assess the severity of scalp psoriasis using the PSSI, which consists of an assessment of erythema, induration, and desquamation on a scale from 0 (none) to 4 (very severe) and the percentage of scalp involved on a scale from 1 (<10% of scalp involved) to 6 (90 to 100% of scalp involved). The composite score is calculated as the sum of the scores for erythema, induration and desquamation multiplied by the score recorded for the extent of scalp area involved. The PSSI ranges from 0 to 72.
Study-S: Percentage of Participants with Achievement of PSS of 0 | Week 16
  The PSS is a 4-item PRO instrument that assesses the severity of psoriasis symptoms in patients with moderate to severe psoriasis, using a recall period of 1 day. The symptoms include pain, redness, itching and burning from psoriasis. Current symptom severity is assessed using a 5-point Likert-type scale ranging from 0 (none) to 4 (very severe).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (38):
- United States (38):
  - Medical Dermatology Specialists /ID# 262915, Phoenix, Arizona
  - Alliance Dermatology and Mohs Center /ID# 255846, Phoenix, Arizona
  - Banner University Medicine Dermatology /ID# 255845, Tucson, Arizona
  - Private Practice - Dr. Tooraj Raoof /ID# 255334, Encino, California
  - Dermatology Research Associates /ID# 255347, Los Angeles, California
  - Clinical Trials Research Institute /ID# 264555, Thousand Oaks, California
  - Florida Academic Dermatology Center /ID# 264065, Coral Gables, Florida
  - Skin Care Research - Hollywood /ID# 255394, Hollywood, Florida
  - GSI Clinical Research, LLC /ID# 255472, Margate, Florida
  - Skin and Cancer Associates, LLP /ID# 255506, Miami, Florida
  - Sullivan Dermatology /ID# 264067, Miami, Florida
  - Renstar Medical Research /ID# 255339, Ocala, Florida
  - Hamilton Research, LLC /ID# 255409, Alpharetta, Georgia
  - Treasure Valley Medical Research /ID# 255671, Boise, Idaho
  - DeNova Research /ID# 264063, Chicago, Illinois
  - Arlington Dermatology /ID# 255330, Rolling Meadows, Illinois
  - The Indiana Clinical Trials Center /ID# 255333, Plainfield, Indiana
  - Dermatology Partners of Leawood /ID# 263244, Leawood, Kansas
  - DermAssociates - Rockville /ID# 263252, Rockville, Maryland
  - Skin Specialists /ID# 262929, Omaha, Nebraska
  - Skin Cancer and Dermatology Institute (SCDI) /ID# 264570, Sparks, Nevada
  - Care Access - Hoboken /ID# 264066, Hoboken, New Jersey
  - Forest Hills Dermatology Group @ Union Turnpike /ID# 255346, Kew Gardens, New York
  - Schweiger Dermatology, P.C. /ID# 255336, New York, New York
  - Darst Dermatology /ID# 255848, Charlotte, North Carolina
  - Wright State Physicians Health Center /ID# 255395, Fairborn, Ohio
  - Apex Clinical Research Center /ID# 263432, Mayfield Heights, Ohio
  - Oregon Dermatology and Research Center /ID# 255670, Portland, Oregon
  - Oregon Medical Research Center /ID# 255332, Portland, Oregon
  - Studies in Dermatology LLC /ID# 262989, Cypress, Texas
  - Modern Research Associates /ID# 263234, Dallas, Texas
  - Center for Clinical Studies - Houston (Binz) /ID# 255396, Houston, Texas
  - U.S. Dermatology Partners Longview /ID# 266325, Longview, Texas
  - Progressive Clinical Research - San Antonio /ID# 263255, San Antonio, Texas
  - Center for Clinical Studies Webster TX /ID# 255518, Webster, Texas
  - Care Access - Danville /ID# 266300, Danville, Virginia
  - Center for Excellence in Dermatology /ID# 264647, Kennewick, Washington
  - North Sound Dermatology /ID# 264565, Mill Creek, Washington

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Song EJ, Ehst B, Glick B, Lewitt GM, Rich P, Ezra N, Bagel J, Anschutz T, Bialik B, Duan C, Ashley D, Patel M, St John G, Setty AR, Ackerman L. Efficacy and Safety of Risankizumab in Genital or Scalp Psoriasis in the UnlIMMited Phase 4 Randomized Clinical Trial at Week 16. Dermatol Ther (Heidelb). 2025 Oct 25. doi: 10.1007/s13555-025-01544-6. Online ahead of print. PMID 41139175
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-702